CLINICAL TRIAL: NCT01363206
Title: GM-CSF and Ipilimumab as Therapy in Metastatic Melanoma, a Phase II Study
Brief Title: Granulocyte Macrophage-Colony Stimulating Factor and Ipilimumab as Therapy in Melanoma
Acronym: GIPI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynn E. Spitler, MD (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Lynn E. Spitler, MD, Director, Northern California Melanoma Center
Organization: Northern California Melanoma Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIPI; BMS 184051 (Other Grant/Funding Number: BMS 184051); Genzyme LEU001 (Other Grant/Funding Number: Genzyme LEU001)
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Malignant Melanoma, Metastatic
Keywords: Melanoma; GM-CSF; Ipilimumab; Immunologic Response
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Colony-Stimulating Factors; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm open label (Experimental): GM-CSF and Ipilimumab
  Interventions: Biological: Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF); Biological: Ipilimumab

INTERVENTIONS:
Biological: Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) — GM-CSF will be administered subcutaneously daily for 14 days in a dose of 125 µg/m2 beginning on D1 of each 21-day cycle for 8 cycles until month 6. Maintenance therapy will begin at month 6 and will consist 14 days of GM-CSF repeated every 3 months for up to 2 years or until disease progression, whichever occurs first.
  Other Names: Leukine; Sargramostim
Biological: Ipilimumab — Patients will be treated with 4 courses of ipilimumab administered every 3 weeks intravenously in a dose of 10 mg/kg, with appropriate stopping/de-escalation rules. Maintenance therapy will begin at month 6 and will consist of ipilimumab in the same dose administered at the end of cycle 4 repeated every 3 months for up to 2 years or until disease progression, whichever occurs first.
  Other Names: Yervoy; Anti-CTLA-4 Monoclonal Antibody

SUMMARY:
The study is an open-label, single arm single Center Phase II study to evaluate the safety and efficacy of the combination of Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF, Leukine) and Ipilimumab (Yervoy) as therapy for patients with unresectable metastatic malignant melanoma.

DETAILED DESCRIPTION:
The study is an open-label, single arm single Center Phase II study to evaluate the safety and efficacy of the combination of Granulocyte Macrophage-Colony Stimulating Factor (GM-CSF, Leukine) and Ipilimumab (Yervoy) as therapy for patients with unresectable metastatic malignant melanoma. The patient sample will be approximately 43 evaluable individuals, males and females 18 years of age or older with measurable metastatic melanoma. Immunologic testing will be done to evaluate correlation with clinical outcome.

Patients will be treated with 4 courses of GM-CSF and ipilimumab administered every 3 weeks. GM-CSF will be administered subcutaneously daily for 14 days in a dose of 125 µg/m2 beginning on D1 of each 21-day cycle. Ipilimumab intravenously in a dose of 10 mg/kg, with appropriate stopping/de-escalation rules. After the initial 3 months (4 cycles) of treatment, GM-CSF administration will continue for 4 additional cycles on the same schedule and dose without ipilimumab for 14 days every 21 days until month 6. Maintenance therapy will begin at month 6 and will consist of ipilimumab in the same dose administered at the end of cycle 4 combined with 14 days of GM-CSF. Administration of this combination will be repeated every 3 months for up to 2 years or until disease progression, whichever occurs first. During the maintenance phase, GM-CSF will only be administered for 14 days in conjunction with ipilimumab and will not be administered in the intervening time period.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, (surgically incurable or unresectable) stage III or IV metastatic malignant melanoma.
2. Prior systemic therapy for metastatic disease is permitted but not required
3. A minimum of 1 measurable lesion according to irRC criteria.
4. ECOG performance status of 0-2.
5. Men and women, age ≥ 18 years.
6. Adequate hematologic, renal and liver function as defined by laboratory values performed within 14 days prior to initiation of dosing.

   * WBC ≥ 2000/uL
   * Absolute neutrophil count (ANC) ≥ 1000/uL
   * Platelet count ≥ 50,000/uL
   * Hemoglobin ≥ 8.0 g/dL
   * Serum creatinine ≤ 3.0 x upper limit of normal
   * Total serum bilirubin ≤ 3.0 x upper limit of normal (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL
   * LDH ≤ 4 times upper limit of laboratory normal
   * Serum aspartate transaminase (ASAT/SGOT) or serum alanine transaminase (ALAT/SGPT) ≤ 2.5 times upper limit of laboratory normal for patients without liver metastases
   * Alkaline phosphatase ≤ 2.5 times upper limit of normal, unless bone metastasis is present in the absence of liver metastases
7. No active or chronic infection with HIV, Hepatitis B, or Hepatitis C
8. Patients must have recovered from effects of major surgery.
9. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 8 weeks after the study in such a manner that the risk of pregnancy is minimized.

WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal. Post-menopausal is defined as:

* Amenorrhea ≥ 12 consecutive months without another cause, or
* For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35mIU/mL].

Exclusion Criteria:

1. Brain metastases that are not treated and not stable for at least 1 month.
2. History of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan.
3. Any other malignancy from which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
4. Autoimmune disease: Patients with a history of inflammatory bowel disease are excluded from this study as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's Granulomatosis), motor neuropathy considered of autoimmune origin (e.g. Guillain-Barré Syndrome).
5. Any underlying medical condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
6. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before trial entry.
7. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab.
8. A history of prior treatment with ipilimumab, CD137 agonist, CTLA-4 inhibitor or agonist; GM-CSF, or monoclonal antibody.
9. Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids.
10. Women of child-bearing potential (WOCBP) who:

    * are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for at least 8 weeks after cessation of study drug, or
    * have a positive pregnancy test at baseline, or
    * are pregnant or breastfeeding
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious) illness
12. Persons of reproductive potential must agree to use and utilize an adequate method of contraception throughout treatment and for at least 8 weeks after study drug is stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Disease control rate at 24 weeks as defined by the immune-related Response Criteria (irRC) | 24 weeks
  Disease control rate will be measured at 24 weeks from the start date of protocol therapy using the immune-related Response Criteria (irRC)

SECONDARY OUTCOMES:
Assessment of immune activation as determined in the Companion Protocol | Three years
  Blood will be drawn for immunologic testing at each patient visit.
Duration of disease control defined as the time from the date of the first treatment dose to the date of first documentation of disease progression as defined by irRC. | Four years
  According to irRC criteria, increase in the size of target lesions or the appearance of new lesions within 12 weeks of the initiation of ipilimumab therapy does not necessarily represent disease progression (as they would using conventional RECIST criteria).
Overall Survival (OS) | Four years
  Overall Survival (OS) is defined as the time from the date of the first treatment dose to date of death due to any cause. In the absence of confirmation of death, survival time will be censored at the last date the patient was known to be alive.
Objective Response Rate (RR) | Two years
  The Objective Response Rate (RR) at any time during the 2 years of study treatment will be evaluated in this study using the immune related Response Criteria (irRC).
Time to Objective response | Three years
  The Time to Objective response is defined as the time from the date of the first treatment dose to the date of first documentation of disease response.
Duration of objective response (CR or PR) | Four years
  The duration of objective response (CR or PR) will be measured from the date the response was first documented to the date of progression or death due to progressive disease, whichever occurs first.
Safety of the combination | Three years
  The safety of the combination as defined by the NCI CTCAE criteria, Version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Spitler, M.D., Principal Investigator — Northern California Melanoma Center, St. Mary's Medical Center
Locations (2):
- United States (2):
  - Northern Californai Melanoma Center, St. Mary's Medical Center, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Spitler LE, Grossbard ML, Ernstoff MS, Silver G, Jacobs M, Hayes FA, Soong SJ. Adjuvant therapy of stage III and IV malignant melanoma using granulocyte-macrophage colony-stimulating factor. J Clin Oncol. 2000 Apr;18(8):1614-21. doi: 10.1200/JCO.2000.18.8.1614. PMID 10764421
- [Background] Hoos A, Eggermont AM, Janetzki S, Hodi FS, Ibrahim R, Anderson A, Humphrey R, Blumenstein B, Old L, Wolchok J. Improved endpoints for cancer immunotherapy trials. J Natl Cancer Inst. 2010 Sep 22;102(18):1388-97. doi: 10.1093/jnci/djq310. Epub 2010 Sep 8. PMID 20826737
- [Background] Kavanagh B, O'Brien S, Lee D, Hou Y, Weinberg V, Rini B, Allison JP, Small EJ, Fong L. CTLA4 blockade expands FoxP3+ regulatory and activated effector CD4+ T cells in a dose-dependent fashion. Blood. 2008 Aug 15;112(4):1175-83. doi: 10.1182/blood-2007-11-125435. Epub 2008 Jun 3. PMID 18523152
- [Derived] Cham J, Zhang L, Kwek S, Paciorek A, He T, Fong G, Oh DY, Fong L. Combination immunotherapy induces distinct T-cell repertoire responses when administered to patients with different malignancies. J Immunother Cancer. 2020 May;8(1):e000368. doi: 10.1136/jitc-2019-000368. PMID 32376721
- See also: This describes the site where the clinical trial is being conducted. — http://www.melanomacenter.com